CLINICAL TRIAL: NCT05011565
Title: The Effects of Hemodynamic, Vascular and Muscular Parameters on Maximal and Submaximal Exercise Capacity in Single-Ventricle Patients With the Fontan Procedure
Brief Title: Hemodynamic, Vascular and Muscular Parameters of Exercise Capacity in Single-Ventricle Patients With Fontan Procedure
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Haluk TEKERLEK, Principal Investigator/Research Assistant, Hacettepe University
Other Study IDs: fontanexercisecapacity
Record Dates: First submitted 2021-07-20; First posted 2021-08-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Single-ventricle; Fontan Procedure; Hemodynamic Instability; Arterial Stiffness; Muscle Oxygenation; Exercise Capacity
MeSH Terms: conditions — Univentricular Heart | interventions — Demography; Muscle Strength

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fontan Group: Fontan Group Inclusion Criteria
  * be between the ages of 8-50
  * Having undergone Fontan operation in our hospital or another center
  * Clinical stability of the patients (preserved ventricular function),
  * No change in ongoing drug therapy that adversely affects clinical stability,
  * At least 1 year after the operation and to be followed in the Pediatric Cardiology Polyclinic of our hospital
  Fontan Group Exclusion Criteria:
  * Inability to access the patient's medical data
  * Neurological and/or genetic musculoskeletal disease
  * Having orthopedic and cognitive problems that prevent testing
  * The patient's and/or family's unwillingness to participate in the study
  Interventions: Other: Demographic and Clinical Characteristics, Maximal Exercise Capacity, Submaximal Exercise Capacity, Hemodynamic Parameters, Muscle Strength, Muscle Oxygenation, Vascular Function
- Control Group: Control Group Inclusion Criteria:
  * Not have cardiovascular, neurological and/or genetic musculoskeletal disease
  * Not having orthopedic and cognitive problems that prevent testing
  * The patient's and/or family's willingness to participate in the study
  Interventions: Other: Demographic and Clinical Characteristics, Maximal Exercise Capacity, Submaximal Exercise Capacity, Hemodynamic Parameters, Muscle Strength, Muscle Oxygenation, Vascular Function

INTERVENTIONS:
Other: Demographic and Clinical Characteristics, Maximal Exercise Capacity, Submaximal Exercise Capacity, Hemodynamic Parameters, Muscle Strength, Muscle Oxygenation, Vascular Function — Demographic and Clinical Characteristics, Maximal Exercise Capacity, Submaximal Exercise Capacity, Hemodynamic Parameters, Muscle Strength, Muscle Oxygenation, Vascular Function

SUMMARY:
After the Fontan procedure applied in patients with a functional or anatomical single ventricle, patients are faced with significant morbidity and mortality risk. Most of the common complications after Fontan such as arrhythmia, cyanosis, ventricular dysfunction, heart failure, atrioventricular valve insufficiency, protein-losing enteropathy, thrombosis, bleeding, venous insufficiency directly or indirectly limit exercise capacity. It has been reported that hemodynamic, vascular and muscular factors may be effective in the decrease of exercise capacity. In previous studies, it has been reported that cardiac output, one of the hemodynamic parameters, is the main factor affecting exercise capacity in patients with Fontan, and this is due to insufficient increase in stroke volume. In addition to the hemodynamic profile, the effects of muscle oxygenation, arterial stiffness and peripheral muscle strength on exercise capacity have been mentioned in different studies. For this reason, it is thought that examining the effects of hemodynamic, vascular and muscular profile together on submaximal and maximal exercise capacity in patients with Fontan will provide information about the mechanisms of influence of different exercise capacities and will provide important information in terms of determining exercise-based rehabilitation programs for such patients.

DETAILED DESCRIPTION:
Fontan operation is a palliative surgical procedure performed in patients with a functional or anatomical single ventricle. After the Fontan procedure, patients face significant risk of morbidity and mortality, and patients with complicated congenital heart disease need to be followed for life by a cardiologist experienced in the care of patients. Annual follow-up is recommended in uncomplicated patients, but more frequent follow-up is required in patients with postoperative complications. Survival rates of 15-20 years after the operation vary between 60-85%. Since there is no ventricular pump to push blood into the pulmonary artery circulation in patients undergoing the Fontan procedure, there is increased systemic venous pressure compared to normal biventricular circulation. Most of the common complications after Fontan are directly or indirectly related to elevation of central venous pressure. These complications include arrhythmia, cyanosis, decreased exercise capacity, ventricular dysfunction, heart failure, atrioventricular valve insufficiency, protein-losing enteropathy, thrombosis, bleeding, venous insufficiency. Patients undergoing the Fontan procedure generally do not experience a normal increase in cardiac output during exercise; therefore exercise capacity is limited. It has been emphasized that hemodynamic, vascular and muscular factors may be effective in decreasing exercise capacity. In previous studies, it has been reported that cardiac output is the main factor affecting exercise capacity in patients with Fontan, and this is due to insufficient increase in stroke volume. However, in previous studies, it has been reported that factors such as insufficient precision of measurements (resting echocardiography in supine position, resting cardiac MRI) and failure to see optimal functions with maximum effort are insufficient to interpret the effects of hemodynamic profile on exercise capacity. Therefore, it is important to evaluate the global and regional myocardial functions in more detail and to determine the hemodynamic profile with speckle tracking echocardiography. In a study, it was reported that atrial tension parameters measured by speckle tracking echocardiography in the Fontan circulation were affected and this was related to functional exercise capacity.. In addition to the hemodynamic profile, the effects of muscle oxygenation, arterial stiffness and peripheral muscle strength on exercise capacity were also mentioned in some separate studies. Changes in muscle oxygenation in children undergoing the Fontan procedure indicate that the balance between the oxygen demand of the tissues and the amount of oxygen supplied is impaired. It is thought that this may be a mechanism that causes a decrease in exercise tolerance in this patient population. Also, the function of peripheral muscles by acting as a pump is particularly important for venous return in the Fontan circulation, and skeletal muscle mass is reduced in patients with Fontan. Studies have shown that leg lean mass is closely related to an increase in blood flow during exercise, and skeletal muscle contractions can generate pulsatile pulmonary blood flow in some patients with Fontan circulation. A relationship was also found between arterial stiffness and cardiorespiratory fitness in pediatric and adult patients with fontan circulation, and it has been reported that practices to increase exercise capacity may be important for the preservation of vascular structures. Exercise capacity in children and adults undergoing the Fontan procedure is evaluated with field tests such as the cardiopulmonary exercise test (CPET) and the 6-minute walk test (6MWT). CPET is very important in terms of providing objective data in terms of cardiopulmonary fitness in the evaluation of maximal exercise capacity and being the gold standard. However, in terms of determining the functional levels of individuals and maintaining their daily living activities, submaximal exercise capacity, which is evaluated with both cheap and practical 6MWT, also gains importance. When the literature was searched, there was no study examining the effects of hemodynamic, vascular and muscular profile on submaximal and maximal exercise capacity. Therefore, in this study, it is aimed to determine and compare the effects of hemodynamics, arterial stiffness and muscle oxygenation on maximal and submaximal exercise capacity in patients with single ventricle who underwent Fontan procedure.

ELIGIBILITY:
Fontan Group Inclusion Criteria

* be between the ages of 8-50
* Having undergone Fontan operation in our hospital or another center
* Clinical stability of the patients (preserved ventricular function),
* No change in ongoing drug therapy that adversely affects clinical stability,
* At least 1 year after the operation and to be followed in the Pediatric Cardiology Polyclinic of our hospital

Fontan Group Exclusion Criteria:

* Inability to access the patient's medical data
* Neurological and/or genetic musculoskeletal disease
* Having orthopedic and cognitive problems that prevent testing
* The patient's and/or family's unwillingness to participate in the study

Control Group Inclusion Criteria:

* Not have cardiovascular, neurological and/or genetic musculoskeletal disease
* Not having orthopedic and cognitive problems that prevent testing
* The patient's and/or family's willingness to participate in the study

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: After obtaining informed consent, control cases will also be evaluated in terms of evaluation parameters within the scope of the study. Patients aged 8-50 years who underwent the fonton procedure and were followed by Hacettepe University, Department of Pediatric Cardiology will be included in the study. A medical and family history, and a physical examination focused on all systems, especially cardiovascular and musculoskeletal systems, will be essential. The eligible patients will be referred to Faculty of Physical Therapy and Rehabilitation after the routine evaluations are completed. Control cases planned to be included in the study to be compared with the results of Fontan patients will be created by inviting the healthy relatives of the patients who applied to our faculty to participate in the study. In addition, control cases will be invited to work through an online advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Maximal O2 consumption | 30-45 minutes
  CPET, the gold standard for cardiorespiratory fitness, will be used in the assessment of maximal exercise capacity based on maximal O2 consumption . Cardiopulmonary exercise test system (Cosmed Quark CPET, Rome, Italy) is a safe method in which the patient can be monitored via ECG during the execution of the individual on a treadmill. The most commonly used method for KPET applied with a treadmill is the Bruce protocol. However, since the Bruce protocol prefers high workload preferences, the Modified Bruce/half Bruce protocol with intermediate increments will be used.
6MWT distance | 15-20 minutes
  Submaximal exercise capacity based on 6MWT distance will be assessed with the 6MWT. The standard test protocol will be applied in a continuous 30 meter corridor. The patient wearing comfortable clothes and shoes will be given standard instructions and verbal guidance during the test. The distance the patient walked during the test will be recorded in meters.
Cardiac output (Q) | 30-45 minutes
  Hemodynamic findings will be evaluated by a specialist doctor with Speckle Tracking Echocardiography. During the evaluation, standard echocardiographic measurements will be performed with transthoracic echocardiography. With these measurements, images suitable for strain analysis will be taken. For the appropriate images taken, deformation analysis will be made using the speckle traking method. The hemodynamic parameters obtained by the analysis will be recorded.
Stroke volume (SV) | 30-45 minutes
  Hemodynamic findings will be evaluated by a specialist doctor with Speckle Tracking Echocardiography. During the evaluation, standard echocardiographic measurements will be performed with transthoracic echocardiography. With these measurements, images suitable for strain analysis will be taken. For the appropriate images taken, deformation analysis will be made using the speckle traking method. The hemodynamic parameters obtained by the analysis will be recorded.
Upper and lower extremity muscle strength | 15-20 minutes
  Upper extremity muscle strength will be measured using a hand grip strength hand dynamometer (Jamar, Sammons Preston, Rolyon, Bolingbrook, IL, USA). Measurements shall be made using standard procedures, right and left sides, with the arms at the side of the trunk, the elbow in a 90 degree flexion position, and the forearm and wrist in a neutral position. The highest of the three measurements will be considered as hand grip strength. For lower extremity muscle strength, the maximum isometric muscle strength of the Quadriceps femoris muscle will be measured with a dynamometer (Lafayette Instrument Company, Lafayette, Indiana).
Muscle oxygen saturation (SmO2) | 30-45 minutes
  Muscle oxygenation will be measured during CPET and 6MWT. Muscle oxygenation will be assessed with the Moxy monitor (Moxy, Fortiori Design LLC, Minnesota, USA), a device that measures local oxygen saturation (SmO2) in muscle capillaries using near infrared spectroscopy (NIRS). During the tests, Moxy will be placed on the vastus lateralis muscle of the participant's dominant leg, midway between the greater trochanter and lateral epicondyle of the femur. After five minutes of sitting resting, SmO2 and THb will be recorded as resting data. During the test, the Moxy data will be recorded continuously and the average value of the recorded data from the beginning to the last moment of the test will be recorded.
Arterial stiffness | 30-45 minutes
  Vascular function will be evaluated using the aortic pulse wave velocity (PWV) technique. During measurement, the Echo probe will be placed in the suprasternal notch, while a pulse Doppler collecting probe will be placed at the Aortic isthmus level and Doppler velocity tracking will be recorded. The time (T1) between the peak of the R wave on the electrocardiogram and the onset of aortic flow on the Doppler will be measured. The Doppler velocity tracking will then be recorded and the time (T2) between the peak R wave (time reference) and the start of the Doppler flow will be measured. T2-T1 is the time between the aortic isthmus of the pulse wave and the accepted point of the abdominal aorta. The distance between the two points (D2 and D1) where the probes are placed will be given by the difference between D2 and D1. PWV will be calculated with the formula D2-D1/T2-T1.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordina R, O'Meagher S, Gould H, Rae C, Kemp G, Pasco JA, Celermajer DS, Singh N. Skeletal muscle abnormalities and exercise capacity in adults with a Fontan circulation. Heart. 2013 Oct;99(20):1530-4. doi: 10.1136/heartjnl-2013-304249. Epub 2013 Jul 11. PMID 23846614
- [Background] Goldstein BH, Urbina EM, Khoury PR, Gao Z, Amos MA, Mays WA, Redington AN, Marino BS. Endothelial Function and Arterial Stiffness Relate to Functional Outcomes in Adolescent and Young Adult Fontan Survivors. J Am Heart Assoc. 2016 Sep 24;5(9):e004258. doi: 10.1161/JAHA.116.004258. PMID 27664807
- [Background] Legendre A, Guillot A, Ladouceur M, Bonnet D. Usefulness of stroke volume monitoring during upright ramp incremental cycle exercise in young patients with Fontan circulation. Int J Cardiol. 2017 Jan 15;227:625-630. doi: 10.1016/j.ijcard.2016.10.087. Epub 2016 Oct 29. PMID 27810293
- [Derived] Tekerlek H, Aykan HH, Vardar-Yagli N, Selcuk SN, Basol-Goksuluk M, Karagoz T, Saglam M. Predictive Role of Atrial Strain, Aortic Stiffness, and Muscle-Related Factors for Maximal and Submaximal Exercise Capacity in Fontan Patients. Pediatr Cardiol. 2025 Dec;46(8):2443-2455. doi: 10.1007/s00246-024-03687-3. Epub 2024 Oct 29. PMID 39470752